CLINICAL TRIAL: NCT07154810
Title: Observational Study to Evaluate Long-term Follow-up of Subjects Implanted With Sustained-release Bimatoprost With the SpyGlass IOL in Subjects With Ocular Hypertension or Mild-to-moderate Open-angle Glaucoma
Brief Title: Observational Study to Evaluate Long Term Outcomes for Ocular Hypertension and Glaucoma Patients Treated With the SpyGlass Bimatoprost Implant System / IOL Combination
Status: Active, not recruiting | Type: Observational
Sponsor: SpyGlass Pharma, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SGP-SPEC-004
Record Dates: First submitted 2025-08-22; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Glaucoma; Cataract; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Cataract; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bimatoprost Implant System / IOL Combination Low Dose
- Bimatoprost Implant System / IOL Combination Medium Dose
- Bimatoprost Implant System / IOL Combination High Dose

SUMMARY:
The goal of this clinical trial is to further observe and learn if the SpyGlass Pharma Bimatoprost Implant System / IOL Combination works to treat cataracts and either ocular hypertension or glaucoma. It will also further observe and learn about the safety of the Bimatoprost Implant System / IOL Combination. The main questions it aims to answer are:

* Does the Bimatoprost Implant System / IOL Combination continue lower the pressure inside the eye to treat ocular hypertension or glaucoma long term?
* Does the Bimatoprost Implant System / IOL Combination continue to correct vision after cataract surgery long term?
* What long term medical problems do participants have when treated with the Bimatoprost Implant System / IOL Combination?

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand a written informed consent and be willing to participate by evidence of signing an informed consent form
* Met all inclusion criteria, participated in and completed the SGP-SPEC-001 study

Exclusion Criteria:

* Planned participation in another clinical trial within 30 days of the initial study visit that, in the investigator's opinion, could confound the study results

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Ocular hypertension or open-angle glaucoma participants in Honduras who completed the SpyGlass Pharma Inc. SGP-SPEC-001 study.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2031-04-14 (Estimated); Study Completion 2031-04-14 (Estimated)

PRIMARY OUTCOMES:
Unmedicated eyes with an IOP Reduction from SGP-SPEC-001 Baseline | From Month 9 post-operative through the end of post-operative follow-up at Month 84
  The proportion of eyes that remain unmedicated and with an IOP reduction ≥ 20% from the SGP-SPEC-001 baseline visit for each follow-up time through the month 84 exam.

OTHER OUTCOMES:
Mean change in unmedicated IOP from SGP-SPEC-001 baseline visit for each follow-up time up to the month 84 exam. | From Month 9 post-operative through the end of post-operative follow-up at Month 84
Number of topical glaucoma medications used in the SGP-SPEC-001 screening for each follow-up time up to the month 84 examination | From Month 9 post-operative through the end of post-operative follow-up at Month 84
Assessment of Postoperative Adverse Events | From Month 9 post-operative through the end of post-operative follow-up at Month 84
Supplementary Safety Parameter - BCDVA | From Month 9 post-operative thorough the end of post-operative follow-up at Month 84
  Best Corrected Distance Visual Acuity (snellen)
Supplementary Safety Parameter - Slit Lamp Examination | From Month 9 post-operative thorough the end of post-operative follow-up at Month 84
  Slit Lamp Examination Findings
Supplementary Safety Parameter - Specular Microscopy | Month 12 post-operative
  Endothelial Cell Density (cells per square millimeter)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Director, Clinical Affairs, Study Chair — SpyGlass Pharma, Inc.
Locations (1):
- Centro Oftalmológico Robles, Santa Rosa de Copán, Honduras

IPD SHARING:
Plan to Share IPD: No
This is an observational extension to a proof of concept trial (first in human).

REFERENCES:
- [Derived] Tan NE, Katz G, Robles M, Gupta PK, Kahook MY, Sussman G, Yoo P, Radcliffe NM. Prospective Pilot Study of Sustained Release Bimatoprost Implant with SpyGlass Intraocular Lens: 3-Year Results. Ophthalmol Ther. 2026 Feb 1. doi: 10.1007/s40123-026-01313-4. Online ahead of print. PMID 41621045